CLINICAL TRIAL: NCT02825186
Title: Dexamethasone (Sterodex) Versus Loteprendol (Lotemax) Eye Drops Following Strabismus Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, MD, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TLV-015-0185
Record Dates: First submitted 2016-05-22; First posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Ophthalmology

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Loteprendol (Experimental): Topical Loteprendol used after strabismus surgery
  Interventions: Drug: Loteprendol etabonate 0.5%
- Dexamethasone (Experimental): Topical Dexamethasone used after strabismus surgery
  Interventions: Drug: Dexamethasone 0.1%

INTERVENTIONS:
Drug: Loteprendol etabonate 0.5% — Steroid eye drops used after strabismus surgery.
  Arms: Loteprendol
Drug: Dexamethasone 0.1%
  Arms: Dexamethasone

SUMMARY:
The purpose of this study is to compare the efficacy and side effects of topical Loteprendol etabonate 0.5% (Lotemax) versus Dexamethasone 0.1% (Sterodex) following strabismus surgery.

DETAILED DESCRIPTION:
This is a randomized prospective study that will involve 100 patients (males and females) undergoing strabismus surgery. All patients will be randomly assigned to receive one of the study drugs (Loteprendol etabonate 0.5% (Lotemax) drops or Dexamethasone 0.1% (Sterodex) drops) after undergoing strabismus surgery. In addition to the study drug all patients (in both groups) will receive topical Ofloxacin 0.3% (Oflox) eye drops. All patients will undergo a complete ophthalmological evaluation before surgery including orthoptic assessment of their strabismus and measurement of intraocular pressure (IOP). Topical treatment with the study drug and topical Ofloxacin 0.3% (Oflox) eye drops will begin on the evening of the surgery, following a schedule that will be the same for both groups: 4 times daily during the first week, 3 times daily for the second group, twice daily for the third week, and as needed for the fourth week. All patients will be examined at 1 day, 1 week, 2 weeks and 4 weeks after surgery by a masked investigator (not the strabismus surgeon).

The parameters to be checked will include:

1. Patient pain and discomfort
2. Conjunctival chemosis
3. Conjunctival hyperaemia
4. Conjunctival discharge
5. Conjunctival gap
6. Intraocular pressure (IOP)
7. Number of pain control medications taken

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing recession strabismus surgery through a fornix approach of one of the horizontal recti muscles (either medial rectus or lateral rectus) or of the inferior oblique muscle
* Must be able to comply with topical treatment
* Must be able to comply with post-operative appointment schedule.

Exclusion criteria:

* Previous ocular surgery (including previous strabismus surgery)
* Ocular pathology
* Family history of glaucoma
* Personal history of allergic drug reaction or allergic conjunctivitis
* More than one muscle operated on
* Adjustable sutures technique
* Patients in whom it is impossible to measure IOP before surgery

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline - Intraocular pressure (IOP) | 1 day before surgery (basline), and 1 day, 1 week, 2 weeks, 4 weeks after surgery
  IOP will be measured by Goldmann applantation tonometry one day before surgery (baseline IOP). In patients in whom Goldmann tonometry is impossible, ICARE tonometer will be used instead. IOP will be measured 1 day, 1 week, 2 weeks, 4 weeks after surgery, at each time point change from baseline IOP will be recorded.
Change from baseline - Conjunctival hyperemia | 1 day before surgery (basline), and 1 day, 1 week, 2 weeks, 4 weeks after surgery
  Conjunctival hyepremia will be measured one day before surgery (basline measurement) using the following scale: 0=no hyperemia, 1=mild (less than one quadrant), 2=moderate (less than half of the conjunctival surface), 3= severe (less than half of the conjunctival surface). Conjunctival hyperemia will be measured 1 day, 1 week, 2 weeks, 4 weeks after surgery, at each time point change from baseline measurement will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel